CLINICAL TRIAL: NCT00762437
Title: A Prospective Clinical Study of Non-Invasive Cooling of Subcutaneous Fat
Brief Title: Non-Invasive Cooling of Fat Cells
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zeltiq Aesthetics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZA07005
Record Dates: First submitted 2008-09-27; First posted 2008-09-30 (Estimated); Results first posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Reduction of Unwanted Fat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment Group (Experimental)
  Interventions: Device: Zeltiq Dermal Cooling Device

INTERVENTIONS:
Device: Zeltiq Dermal Cooling Device — Non-invasive cooling is applied to the treatment area with a defined cooling rate and duration.

SUMMARY:
The purpose of this study is to evaluate a non-invasive cooling device to determine if cold exposure will consistently result in a reduction of subcutaneous fat.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects > 18 years of age.
2. Subject has clearly visible fat on an area of the body appropriate for treatment with the non-invasive Zeltiq cooling device such as the flanks, thighs, abdomen or back.
3. Subject has not had weight change fluctuations exceeding 10 pounds in the preceding month and plans to maintain their weight to within ±10 pounds over the next 6 months.
4. Subject has read and signed a written informed consent form.

Exclusion Criteria:

1. Subject has had liposuction, or another surgical procedure(s) or mesotherapy in area of intended treatment within the past 2 years.
2. Subject has a known history of subcutaneous injections into the area of intended treatment (e.g., cortisone) within the past 6 months.
3. Subject has a known history of cryoglobulinemia, cold urticaria, or paroxysmal cold hemoglobinuria.
4. Subject has used diet pills within the past 6 months.
5. Subject is unable or unwilling to comply with the study requirements.
6. Subject has any dermatological conditions or scars within the location of the test sites that may interfere with the treatment or evaluation.
7. Subject is currently enrolled in a clinical study of any other unapproved investigational drug or device.
8. Patient is pregnant or intending to become pregnant in the next 9 months.
9. Patient is lactating or has been lactating in the past 9 months.
10. Any other condition or laboratory value that would, in the professional opinion of the investigator, potentially affect response or participation in this clinical study, or would pose an unacceptable risk to the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2008-01; Primary Completion 2009-11-17 (Actual); Study Completion 2009-12-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Investigational Site, Sacramento, California
  - Investigational Site, San Diego, California
  - Investigational Site, Washington D.C., District of Columbia
  - Investigational Site, Miami, Florida
  - Investigational Site, Chicago, Illinois
  - Investigational Site, Baltimore, Maryland
  - Investigational Site, Boston, Massachusetts
  - Investigational Site, Minneapolis, Minnesota
  - Investigational Site, Hackensack, New Jersey
  - Investigational Site, New York, New York
  - Investigational Site, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: Non-invasive cooling was applied to the treatment area with a defined cooling rate and duration.
Period: Overall Study
Arm/Group | All Participants
Started | 175
Completed | 156
Not Completed | 19
Not completed — Lost to Follow-up | 7
Not completed — Missed final study visit | 11
Not completed — No treatment (unable to attach sleeve to participant) | 1

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Zeltiq Dermal Cooling Device: Non-invasive cooling was applied to the treatment area with a defined cooling rate and duration.
Arm/Group | All Participants
Number analyzed (Participants) | 175
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.9 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 132
  Male | 43

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Visible Improvement in Treated Area
Description: Investigator assessment to document any visible improvement in the treatment area.
Time Frame: 4 months
Population: Participants with evaluable data for each body site were included in this analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Back Fat; Love Handles: Non-invasive cooling was applied to the treatment area with a defined cooling rate and duration.
Arm/Group | Back Fat | Love Handles
Number analyzed (Participants) | 69 | 58
percentage of participants | 65.2 [52.8 to 76.3] | 82.8 [70.6 to 91.4]

2. Secondary Outcome: Participant Satisfaction
Description: Percentage satisfaction with the Zeltiq procedure as determined by the results of a subjects satisfaction questionnaire.
Time Frame: 4 months
Population: Participants with evaluable data for each body site were included in this analysis. The row titled "Percentage of participants 'Both Satisfied and Dissatisfied' on Subject Satisfaction Questionnaire" was not applicable to the Love Handle treatment area, so no data were collected.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Back Fat | Love Handles
Number analyzed (Participants) | 74 | 65
percentage of participants
  Percentage of participants with "overall satisfaction" on Subject Satisfaction Questionnaire | 51.4 [39.4 to 63.1] | 58.5 [45.6 to 70.6]
  Percentage of participants "Dissatisfied" on Subject Satisfaction Questionnaire | 8.1 [3.0 to 16.8] | 6.2 [1.7 to 15.0]
  Percentage of participants "Neither Satisfied nor Dissatisfied"on Subject Satisfaction Questionnaire | 32.4 [22.0 to 44.3] | 35.4 [23.9 to 48.2]
  Percentage of participants "Both Satisfied and Dissatisfied" on Subject Satisfaction Questionnaire: number analyzed (Participants) | 74 | 0
  Percentage of participants "Both Satisfied and Dissatisfied" on Subject Satisfaction Questionnaire | 8.1 [3.0 to 16.8] |

ADVERSE EVENTS:
Time Frame: All-cause mortality and adverse event tables include events reported from first treatment through study completion, an average of 6 months.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/175
Serious Adverse Events (participants affected / at risk) | 0/175
Other Adverse Events (participants affected / at risk) | 12/175
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=175)
Syncope (Cardiac disorders) | 2
Fainting (Vascular disorders) | 1
Chest Pain (General disorders) | 1
Elevated Heart Rate (Cardiac disorders) | 1
Hyperlipidemia (Metabolism and nutrition disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Vasovagal event (General disorders) | 2
Gallbladder attack (Hepatobiliary disorders) | 1
Toe Pain (General disorders) | 1
Tingling (Nervous system disorders) | 1
Itching (Skin and subcutaneous tissue disorders) | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1
Rib Soreness (General disorders) | 1
(General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.